CLINICAL TRIAL: NCT03228771
Title: Socket Augmentation Using Atorvastatin With Or Without PRGF Derived Fibrin Scaffold (Clinical and Histomorphometric Study)
Brief Title: Socket Augmentation Using Atorvastatin With Or Without PRGF (Clinical and Histomorphometric Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha Nasr, Researcher, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RECM041515
Record Dates: First submitted 2015-05-26; First posted 2017-07-25 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Socket Preservation
Keywords: PRGF; Statins; socket augmentation
MeSH Terms: interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Intervention Model Description: 3 Groups: Group 1: statin loaded in PRGF Group 2: statin loaded in methylcellulose gel Group 3: control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PRGF/ATV (Active Comparator): Group I (PRGF/ATV) : It was included 10 patients undergoing single tooth extraction followed by socket fill with 1.2% Atorvastatin loaded in PRGF derived fibrin scaffold then suturing the socket. All patients will receive implants after taking the bone biopsy after 8 weeks for histomorphometric analysis.
  Intervention: Atorvastatin drug loaded in platelets rich in growth factors (PRGF).
  Interventions: Drug: PRGF/ATV
- ATV gel (Active Comparator): Group II (ATV gel) : Will include 10 patients undergoing single tooth extraction followed by socket fill with 1.2% Atorvastatin in methyl cellulose gel then suturing the socket. All patients will receive implants after taking the bone biopsy after 8 weeks for histomorphometric analysis.
  Interventions: Drug: ATV gel
- Empty socket (No Intervention): Group III Empty socket( control) : Will include 10 patients undergoing single tooth extraction then suturing the socket. All patients will receive implants after taking the bone biopsy after 8 weeks for histomorphometric analysis.

INTERVENTIONS:
Drug: PRGF/ATV — Atorvastatin loaded in PRGF fibrin scaffold
  Other Names: platelets rich in growth factors
  Arms: PRGF/ATV
Drug: ATV gel — Atorvastatin loaded in methyl cellulose gel
  Other Names: Atorvastatin gel
  Arms: ATV gel

SUMMARY:
Despite the numerous studies describing the benefits of PRGF (plasma rich in growth factors) and Statins separately , there has been a lack of clinical investigation into the simultaneous use of these agents in socket augmentation. Therefore the main objective of this study is to evaluate socket bone dimensions and quality following the use of PRGF derived fibrin scaffold as a carrier for Atorvastatin in socket augmentation clinically and histomorphometrically.

DETAILED DESCRIPTION:
Despite the numerous studies describing the benefits of PRGF (plasma rich in growth factors) and Statins separately , there has been a lack of clinical investigation into the simultaneous use of these agents in socket augmentation.

Plasma Rich in Growth Factors (PRGF) have given rise to an optimized and safer product rich in growth factors which might be essential to proper tissue repair and wound healing. PRGF acts on already differentiated cells, such as preosteoblasts and osteoblasts. However , they do not exert any effects on the stem cells present in bone tissue, whose differentiation is regulated by bone morphogenetic proteins (BMPs). Some pharmacologic compounds could offer a safe and cost effective alternative to this problem and can affect bone regeneration. Statins are widely used group of cholesterol lowering drugs that act on the mevalonate pathway by being a competitive inhibitors of the rate limiting enzyme 3-hydroxy-3-methylglutaryl coenzyme A (CoA) reductase (HMG-CoA reductase). Statins increase normal bone formation by promoting osteoblast proliferation and differentiation and protecting the osteoblasts from apoptosis. In addition, they reduce osteoclastogenesis by inhibiting osteoclastic differentiation. Statins increase BMP-2 gene expression and subsequently promote bone formation.This study hypothesized that use of PRGF fibrin scaffold in socket preservation owing to its biocompatibility, ease of use, stimulation of production of growth factors and its effect on the already differentiated osteoblasts, when combined with statin with its effect on progenitor stem-cells could stimulate the differentiation of stem cells to osteoblasts, prevent bone resorption and stimulate bone formation at the extraction socket. Therefore the main objective of this study is to evaluate socket bone dimensions and quality following the use of PRGF derived fibrin scaffold as a carrier for Atorvastatin in socket augmentation clinically and histomorphometrically.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients as evidenced by Burkett's oral medicine health history questionnaire.
* Both sexes.
* Age from 20 - 50 years old.
* Having at least one hopeless tooth indicated for extraction.
* Patient should agree to sign a written consent after the nature of the study will be explained.

Exclusion Criteria:

* Smokers.
* Pregnant and breast feeding females.
* Prisoners and handicapped patients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
clinical measurements Ridge width | 1 year
  Ridge width

SECONDARY OUTCOMES:
clinical measurements ridge height | 1 year
  Ridge height

OTHER OUTCOMES:
histomorphometric analysis | 1 year
  Bone core biopsy for histomorphometric analysis to measure osteoid tissues and mineralized bone

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Ghaffar, Professor, Study Director — Ain Shams University; Ola M Ezzatt, Lecturer, Study Chair — Ain Shams University
Locations (1):
- Faculty of dentistry-Ain shams University, Cairo, Egypt

DOCUMENTS (3):
  • Study Protocol (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03228771/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03228771/SAP_001.pdf
  • Statistical Analysis Plan (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03228771/SAP_002.pdf